CLINICAL TRIAL: NCT04196023
Title: Ca:Mg Ratio and Cognitive Function in the Personalized Prevention of Colorectal Cancer Trial
Brief Title: Ca:Mg Ratio and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Qi Dai, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 100106a; R01CA149633 (NIH); R01CA202936 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Function
MeSH Terms: interventions — magnesium diglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium treatment (Active Comparator): Participants will be assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate; Dietary Supplement: Placebo
- placebo (Placebo Comparator): Participants will be assigned to placebo group
  Interventions: Dietary Supplement: Magnesium glycinate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Oral administration of magnesium glycinate daily for 12 weeks
Dietary Supplement: Placebo — Oral administration of identical-appearing placebo daily for 12 weeks

SUMMARY:
Between 2000 and 2015, mortality due to Alzheimer's disease (AD) increased by 123%. No drugs have yet been approved to stop or slow the progression of AD. A delay of five years in the expression of AD would reduce the incidence rate by half. Thus, it is critical to develop novel prevention strategies to delay the onset of this common disease.

As an ancillary study conducted within a precision-based randomized trial (R01CA149633; PI, Dai & Yu]"), the investigators reduced Ca:Mg ratios to 2.3 through 3-month personalized Mg supplementation among those who consumed high Ca:Mg ratio diet, but otherwise in good general health. The investigators test the hypothesis that actively reducing the Ca:Mg ratio among those aged >65 years who consume high Ca:Mg ratio diets improves cognitive function compared to the placebo arm. The investigators further conduct molecular epidemiologic studies to understand the molecular mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from our parent study (Personalized Prevention of Colorectal Cancer Trial, NCT#01105169, IRB#100106);
2. Participants who completed the MoCA

Exclusion Criteria:

1. Participants did not provide their blood samples in the parent study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

REFERENCES:
- [Background] Zhu X, Borenstein AR, Zheng Y, Zhang W, Seidner DL, Ness R, Murff HJ, Li B, Shrubsole MJ, Yu C, Hou L, Dai Q. Ca:Mg Ratio, APOE Cytosine Modifications, and Cognitive Function: Results from a Randomized Trial. J Alzheimers Dis. 2020;75(1):85-98. doi: 10.3233/JAD-191223. PMID 32280092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants, aged 40-85 y, with colorectal polyp or polyp-free individuals with high risk of colorectal cancer and had a calcium intake of ≥700 and <2000 mg/d, and their calcium-to-magnesium intake ratio was >2.6 (based on baseline two 24-hour dietary recalls) and completed MoCA assessment were recruited from Vanderbilt patient sources from Dec. 12, 2012 to Jan 30, 2016.
Groups:
- Participants Were Assigned to Magnesium Glycinate: Magnesium glycinate: Oral administration of magnesium glycinate daily for 12 weeks
- Participants Were Assigned to Placebo: Placebo: Oral administration of identical-appearing placebo daily for 12 weeks
Period: Overall Study
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
Started | 62 | 67
Completed | 59 | 64
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Will be Assigned to Magnesium Glycinate: Magnesium glycinate: Oral administration of magnesium glycinate daily for 12 weeks
- Participants Will be Assigned to Placebo: Placebo: Oral administration of identical-appearing placebo daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Participants Will be Assigned to Magnesium Glycinate | Participants Will be Assigned to Placebo | Total
Number analyzed (Participants) | 62 | 67 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 91
  >=65 years | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.7) | 61.2 (8.0) | 60.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 28 | 29 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 60 | 66 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 67 | 129
Overall MoCA Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Cognitive function was measured by the Montreal Cognitive Assessment (MoCA) which is used to evaluate people with memory loss or other symptoms of cognitive decline. Scores on the MoCA range 0-30. Higher values represent a better outcome. A score of 26 or above is considered normal.
  units on a scale | 27.0 (2.7) | 27.2 (2.2) | 27.1 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Overall Score Changes From Baseline by Magnesium Treatment vs. Placebo
Description: Montreal Cognitive Assessment (MoCA) Scoring: The test consists of 30 items, and each item is worth one point, resulting in a maximum score of 30. A higher score indicates better cognitive functioning.
  The changes of MoCA score=Score at 12 weeks minus Score at baseline.
Time Frame: 12 weeks
Population: IRB approval was obtained to add the MoCA component on Dec.11 2012. From Dec. 12, 2012 to Jan 30, 2016, 129 participants enrolled the study. Among them, 123 (95.3%) completed pre-and post- treatment MoCA were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
Number analyzed (Participants) | 59 | 64
score on a scale | 1.1 (2.3) | 0.6 (2.6)
Statistical Analysis 1: Comparison: Participants Were Assigned to Magnesium Glycinate vs Participants Were Assigned to Placebo; Test type: Superiority; p = 0.20, general linear model — p-value was calculated using GLM. Statistical significance was determined using an alpha level of 0.05; adjusted for age, sex, education and baseline overall MoCA score

2. Primary Outcome: Overall Score Changes From Baseline by Magnesium Treatment vs. Placebo (Aged ≤65 Years Old)
Description: as for outcome 1
Time Frame: 12 weeks
Population: 123 participants who completed both pre- and post-treatment MoCA tests are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
Number analyzed (Participants) | 44 | 49
score on a scale | 0.7 (2.0) | 0.6 (2.8)
Statistical Analysis 1: Comparison: Participants Were Assigned to Magnesium Glycinate vs Participants Were Assigned to Placebo; Test type: Superiority; p = 0.90, general linear model — p-value was calculated using GLM model. Statistical significance was determined using an alpha level of 0.05; GLM model additionally adjusting for age, sex, education and baseline level

3. Primary Outcome: Overall Score Changes From Baseline by Magnesium Treatment vs. Placebo (Aged >65 Years Old)
Description: as for outcome 1
Time Frame: 12 weeks
Population: 123 participants who completed pre-and post- treatment MoCA were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 2.3 (2.7) | 0.5 (1.9)
Statistical Analysis 1: Comparison: Participants Were Assigned to Magnesium Glycinate vs Participants Were Assigned to Placebo; Test type: Superiority; p = 0.01, general linear model — p-value was calculated using GLM model. Statistical significance was determined using an alpha level of 0.05; GLM model additionally adjusting for age, sex, education and baseline level

4. Primary Outcome: Changes From Baseline of 5-mC Methylation (CpG Sites) in Apolipoprotein E (APOE) by Magnesium Treatment vs. Placebo
Description: 5-mC methylation (CpG sites) in Apolipoprotein E (APOE) were measure by TET-assisted bisulfite (TAB)-Array.
  5-mC methylation changes=value at 12 weeks minus value at baseline.
Time Frame: 12 weeks
Population: 123 participants who completed both pre- and post-treatment MoCA tests were included in the analysis.
Measure: Mean (Standard Deviation); unit: CpG sites
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
Number analyzed (Participants) | 59 | 64
CpG sites
  cg18768621 | 0.006 (0.025) | -0.003 (0.025)
  cg13496662 | -0.018 (0.060) | 0.006 (0.067)
Statistical Analysis 1: Comparison: Participants Were Assigned to Magnesium Glycinate vs Participants Were Assigned to Placebo; Test type: Superiority; p = 0.05, general linear model — p-value was calculated using GLM model and false discovery rate (FDR)-adjustment. Statistical significance was determined using an alpha level of 0.05; GLM model additionally adjusting for age, sex, education and baseline level

ADVERSE EVENTS:
Time Frame: In the 12 weeks trial, we conducted safety and compliance calls to collect adverse event data.
Description: The definition of adverse event and/or serious adverse event is from the clinicaltrials.gov Definitions.
  We conducted safety and compliance calls to collect adverse event data.
Arm/Group | Participants Were Assigned to Magnesium Glycinate | Participants Were Assigned to Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/67
Other Adverse Events (participants affected / at risk) | 4/62 | 2/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Were Assigned to Magnesium Glycinate (N=62) | Participants Were Assigned to Placebo (N=67)
some bleeding after the rectal biopsy procedure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — abdominal pain
may interact with blood pressure medication (Vascular disorders) | 1 (1) | 0 (0)
weight gain, migraine and swelling with arthritic pain in fingers (General disorders) | 1 (1) | 0 (0)
feel sick (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04196023/Prot_SAP_000.pdf